CLINICAL TRIAL: NCT00700128
Title: Prevention of Menstrual Migraines: Effects of Continuous Oral Contraceptives to Combination With Prophylactic Frovatriptan Use During Hormone Free Intervals
Brief Title: Prevention of Menstrual Migraines: Using Frovatriptan or Placebo During Hormone Free Intervals
Acronym: MAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scott and White Hospital & Clinic (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Patricia Sulak, MD prinicipal investigator, Scott and White Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 060714
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Migraines; Bleeding; Spotting
Keywords: headaches; migraines; breakthrough bleeding; breakthrough spotting; menstrually associated migraines; breakthrough bleeding or breakthrough spotting
MeSH Terms: conditions — Migraine Disorders; Hemorrhage; Metrorrhagia; Headache | interventions — frovatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2 (Experimental): Frovatriptan or placebo given in a certain sequence depending on what group that the woman are randomized to.
  Interventions: Drug: frovatriptan; Drug: placebo
- Group1 (Experimental): Group I will receive in a different sequence either frovatriptan 2.5 mg or placebo bid starting the last day of taking OC and continuing during the hormone free interval (HFI) of 4 days.
  Interventions: Drug: frovatriptan; Drug: placebo

INTERVENTIONS:
Drug: frovatriptan — Frovatriptan 2.5 mg or placebo given Bid starting on the last day of OC before taking the 4 day HFI. They will take a total of 10 pills max per HFI.
  Other Names: frova
  Arms: Group 2
Drug: frovatriptan — frovatriptan 2.5 mg bid or placebo starting on the last day of OC and continuing during the 4 day HFI.
  Other Names: frova
  Arms: Group1
Drug: placebo — placebo

SUMMARY:
This study will examine the combined effects of a continuous oral contraceptive (OC) regimen with supplemental frovatriptan therapy on headache severity and occurrence in subjects with documented Menstrually Associated Migraines (MAM). The subjects enrolling in the study will have cyclic menses either due to spontaneous ovulation or use of cyclic hormonal contraception (pill, patch, or ring). Enrolled subjects will start a continuous OC regimen following two baseline menstrual cycles. If breakthrough bleeding/spotting (BTB/BTS) occurs, the subject will institute a 4-day hormone-free interval (HFI). In an attempt to prevent/lessen the severity of headache during the HFI, subjects will be randomized to prophylactic administration of a triptan or placebo during this period. If no BTB/BTS occurs after 80 days of continuous pills, the subject will institute a 4-day HFI during which they will be randomized into triptan or placebo groups.

The purpose of this research study is to examine the effects of continuous oral contraceptive pills and frovatriptan on headaches that occur around the time of your period. Many woman take continuous oral contraceptive pills (OC) and when OCs are stopped they may get headaches. This study will look if taking frovatriptan around the time of the period will affect the headache, and how it will be affected. Frovatriptan is an FDA approved drug for migraine headaches.

This study is a prospective pilot trial.The study will last approximately 35-39 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Woman may be on birth control pill (OC), patch or NuvaringTM (vaginal ring) taken in the traditional 21/7 or 24/4 manner, which means ever month they have a period. If they are taking it continuously (without a period), you must be willing to take your birth control 24/4 (4 days taking hormone free interval, HFI) for 2 months.
* If you are not on OCs, patch or NuvaringTM you must have a period every 21-40 days.
* You must not want to get pregnant for 12 months.
* Women have headaches around the time of their period.

Exclusion Criteria:

* BMI > 38
* If you smoke and are age 35 years old or greater or if are under 35 years old and smoke over 10 cigarettes a day
* If you have or had an aura with your headaches (An aura is a temporary sensation, like bright lights that come before you experience the headache.)
* Headaches are not occurring during the time of your period.
* Blood Pressure > 140/90 or you take more than a single antihypertensive medication (excluding diuretics) and are age 40 or greater.
* Contraindications to combination estrogen/progestin hormonal contraception.
* Desire to become pregnant in the next 12 months.
* Refuse to avoid any ergot-based medication, triptan medication or isometheptene/midrin during their hormone free interval or the one day before the hormone free interval
* Stroke
* Breast Cancer
* Blood clots in your legs, lung or anywhere else in your body
* Diabetes mellitus
* Heart attack
* Liver disease
* Lupus Erythematosus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Comparing baseline menstrually associated migraines (MAMs)to headache occurrence and severity after the implementation of continuous OC therapy. | 24 weeks

SECONDARY OUTCOMES:
Compare amount of bleeding and spotting within subjects in relation to duration of extended oral contraceptive pills (OCP) use for those previously using the 21/7 day regimen and those initiating OCP use directly from spontaneous cycling. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Sulak, MD, Principal Investigator — Scott and White Hospital
Locations (1):
- Scott & White Memorial Hospital, Temple, Texas, United States

REFERENCES:
- [Background] 1. Lipton RB, Bigal ME, Diamond M, Freitag F, Reed ML, Stewart WF; AMPP Advisory Group. Migraine prevalence, disease burden, and the need for preventive therapy. Neurology 2007; 68(5):343-9. 2. Tozer BS, Boatwright EA, David PS, Verma DP, Blair JE, Mayer AP, Files JA. Prevention of migraine in women throughout the life span. Mayo Clin Proc. 2006;81(8):1086-91. 3. Macgregor EA. Menstrual migraine: a clinical review. Journal of family planning and reproductive health care, 2007. 33(1), 36-47. 4. Brandes JL. The influence of estrogen on migraine: a systematic review. JAMA, 2006; 295(15):1824-30. 5. Sulak PJ, Scow RD, Preece C, Riggs MW, Kuehl TJ. Hormone withdrawal symptoms in oral contraceptive users. Obstet Gynecol 2000; 95:261-6. Sulak P, Willis S, Kuehl T, Coffee A, Clark J. Headaches and oral contraceptives: impact of eliminating the standard 7-day placebo interval. Headache. 2007;
- See also: Scott & White Memorial Hospital Clinical Trials — http://www.sw.org/web/SW/researchAndEducation/iwcontent/public/research/en_us/html/research_clinicaltrials_clinicaltrials.html#Obstetrics_Gynecology